CLINICAL TRIAL: NCT00167050
Title: The Pathogenesis of Superior Limbic Keratoconjunctivitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700634
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2005-06

CONDITIONS: Superior Limbic Keratoconjunctivitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Superior limbic keratoconjunctivitis (SLK) was first described in detail as a clinical entity by Frederick Theodore in 1963. The clinical picture of SLK is well documented, but the etiology is still unknown. This project will be conducted into through two parts: one is to investigate the presentation of chemokine receptors on mast cell and matrix metalloproteinases on fibroblasts by immunohistochemistry method from the pathological specimens of SLK patients who received conjunctiva resection as the treatment. The other part is to investigate the mRNA level of those chemokine receptors via reverse transcription - polymerase chain reaction from the conjunctiva collecting form SLK patients.

DETAILED DESCRIPTION:
1. Specimens collection:

   We will collect the specimens in two different parts. One part is to collect all the paraffinized block of the SLK patients to get fifteen copies of 5-μm section of each paraffinized block from the Department of Pathology. All the slides will be deparaffinized and rehydration for further immunohistochemistry (IHC) stain . Primary antibodies for IHC stain include chemokine receptors (CXCR1, CXCR2, CXCR3, CXCR4, CCR1. CCR3, CCR4, CCR5, CD30L) and matrix metalloproteinases (MMP-1, -2, -3, -9).

   Another part of this study is to collect the conjunctiva of SLK patients and normal control patients. This part of the clinical study is sent for IRB approval concomitantly. We will collect the conjunctiva of SLK patients when they receive conjunctival resection as the treatment in the following one year. And the normal control conjunctiva will be obtained while the patients come to our hospital for cataract surgery or retinal surgery with redundant conjunctiva noted after peritomy. The fresh conjunctiva will be stored in -80℃ before RNA isolation. All the tissue will be processed into RNA and reverse transcripted into cDNA. Polymerase chain reaction will be done with the primers, including CXCR1, CXCR2, CXCR3, CXCR4, CCR1, CCR3, CCR4, CCR5, and CD30L.
2. Preparation of RNA and cDNA:

   Total RNA will be extracted from the conjunctiva of SLK and control groups with Trizol reagent (Life, Gaithersburg, MD, USA). One microgram of total RNA from each sample will be annealed for 5 min at 70℃ with 500 ng oligo(dT) (Fermentas, Hanover, MD, USA) and reverse transcribed to cDNA by 200u RevertAid™ M-MuLV Reverse Transcriptase (Fermentas, Hanover, MD, USA) per 20 µl reaction for 1 hr at 42℃. The reaction will be stopped by heating for 10 min at 70℃.
3. Polymerase chain reaction (PCR):

   PCR will be performed on the resultant cDNA from each sample with specific primers for human chemokines, chemokine receptors and glyceraldehydes-3-phosphate dehydrogenase (GAPDH). The amplification will be performed with a thermocycler. The 25-μl reaction mixture consists of 2 μl cDNA, 1 μl sense and antisense primer, 12.5 μl 2x PCR mix. Conditions for amplifying each chemokine and chemokine receptor are as follows: denaturation, 1 min at 94℃, and elongation, 3 min at 72℃. The annealing temperature and the cycle of annealing for chemokines and chemokine receptors will fit the requested temperature and the appropriate number of annealing cycles of each specific primer. At the end of amplification, the reaction mixture will be heated for 10 min at 72℃ and then cooled to 4℃. A 10-μl sample of each PCR product will be separated by performing gel electrophoresis on 2% agarose containing ethidium bromide (Sigma, St Louis, MO, USA). The 2% agarose gel will be analyzed under ultraviolet light against the DNA molecular length markers. The internal control of each sample is human GAPDH.
4. Immunohistocytometry (IHC):

A pre-determined optimal dilution of the primary antibody specifically against mast cell tryptase, associated chemokines, chemokine receptors, MMPs, and inflammatory cytokines will be used for IHC. All IHC staining will be performed at room temperature. Sections are then deparaffinized in xylene and made hydrophilic by immersion in a graded series of ethanol dilutions (100, 95, 80, and 60%). All slides are immersed in antigen retrieval solution (Dako ,S3307, SA, USA) and autoclaved for 10 min. Sections are quenched with 3% fresh H2O2 for 10 min to inhibit endogenous tissue peroxidase activity that might interfere with the result of staining, and rinsed with 1x PBS for 5 min twice. Sections are further incubated in blocking serum solution for 30 min and then incubated at 37℃ for 1 h with primary antibody in a humid chamber. After washing with 1x PBS for 5 min twice, the sections are then incubated with biotinylated secondary antibody solution for 30 min. The horseradish peroxidase-conjugated streptavidin-biotin complex is subsequently spread evenly over the sections and incubated for 30 min. The sections are washed with 1x PBS for 5 min twice, then incubated with diaminobenzidine (DAB) perioxidase substrate solution for 15 min followed by wash with 1x PBS. Finally, the section are counterstained with an adequate volume of hematoxylin, and then mounted.

ELIGIBILITY:
Inclusion Criteria:

* Superior limbic keratoconjunctivitis patients who receive conjunctiva resection

Exclusion Criteria:

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-07; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Sun YC, Hsiao CH, Chen WL, Hu FR. Overexpression of matrix metalloproteinase-1 (MMP-1) and MMP-3 in superior limbic keratoconjunctivitis. Invest Ophthalmol Vis Sci. 2011 Jun 1;52(6):3701-5. doi: 10.1167/iovs.10-6324. PMID 21357403
- [Derived] Sun YC, Hsiao CH, Chen WL, Wang IJ, Hou YC, Hu FR. Conjunctival resection combined with tenon layer excision and the involvement of mast cells in superior limbic keratoconjunctivitis. Am J Ophthalmol. 2008 Mar;145(3):445-452. doi: 10.1016/j.ajo.2007.10.025. Epub 2008 Jan 16. PMID 18201682